CLINICAL TRIAL: NCT03081416
Title: "THINK Trial: Treatment of Headache With IntraNasal Ketamine: A Randomized Controlled Trial Evaluating the Efficacy of Intranasal Ketamine Versus Standard Therapy in the Management of Primary Headache Syndromes in the Emergency Department"
Acronym: THINK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Danny Villalobos, Nellis AFB Deputy Flight Commander, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.2016.072
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-03

CONDITIONS: Headache; Intranasal Ketamine
MeSH Terms: conditions — Headache | interventions — Ketamine; Saline Solution; Metoclopramide; Standard of Care; Ketorolac; Dexamethasone; Diphenhydramine

STUDY DESIGN:
Intervention Model Description: Two arm-Randomized placebo controlled
Who Masked: Participant
Masking Description: Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intranasal Ketamine arm (Experimental): Intranasal ketamine administered to participant
  Interventions: Drug: Ketamine; Drug: Normal saline
- Standard Therapy (Active Comparator): Reglan 10 mg; Benadryl 25 mg administered to all participants Toradol 15-30 mg; dexamethasone 10 mg added at treating providers discretion.
  Interventions: Drug: Metoclopramide; Drug: Ketorolac; Drug: Dexamethasone; Drug: Benadryl

INTERVENTIONS:
Drug: Ketamine — Intranasal ketamine administration
  Arms: Intranasal Ketamine arm
Drug: Normal saline
  Other Names: Placebo
  Arms: Intranasal Ketamine arm
Drug: Metoclopramide — Standard therapy
  Other Names: Standard therapy
  Arms: Standard Therapy
Drug: Ketorolac — standard therapy
  Arms: Standard Therapy
Drug: Dexamethasone — Standard therapy
  Arms: Standard Therapy
Drug: Benadryl — Standard therapy
  Arms: Standard Therapy

SUMMARY:
This is a randomized, single-blind, placebo controlled trial to evaluate the efficacy of sub-dissociative dose ketamine versus standard care therapy for acute headache management of in patients presenting to the emergency department with headache as the chief compliant.

DETAILED DESCRIPTION:
This is a randomized, single-blind, placebo controlled trial to evaluate the efficacy of sub-dissociative dose ketamine versus standard care therapy for acute headache management of in patients presenting to the emergency department with headache as the chief compliant. Standard care will include 25 mg of diphenhydramine (DIP) IV, 10 mg of metoclopramide (MET) IV, +/- 15-30 mg ketorolac and +/- 10 mg of dexamethasone (DEX) IV the discretion of the treating provider. This study has been approved by Brooke Army Medical Center (BAMC) institutional review board and clinicaltrials.gov registration is pending.

A convenience sample of patients 18 to 65 years of age with a chief complaint of headache will be considered for enrollment. Potential subjects are those presenting to the SAMMC ED with a chief complaint of headache. Attempts to engage subjects earlier in their ED Course (EDC) will be made. This will mitigate interruptions in the subject's EDC, possible withdrawals from the control group, and lack of subject interest in the study. The triage nurse will inform the PI or AI of any patient presenting to the ED with a chief complaint of headache. Patients meeting inclusion criteria will be provided with a brochure briefing them on the study. If they are willing to participate, then a member of the research team will obtain written consent.

Patient screening, enrollment, patient consents, and data collection will be performed by the PI or AI. Each AI will complete training regarding study details, inclusion/exclusion criteria, atomization, intranasal delivery, and ketamine pharmacokinetics which will be conducted by the PI.

Once a patient is consented the team member will obtain a study packet, and the patient will be assigned a study identification number. The study packet will contain the required forms, surveys, Wand documentation forms. The study personnel will then write on the patient's standard order sheet "SDDK Protocol, Patent #__, __kg"

All females of child-bearing age that have not had a hysterectomy or tubal ligation will receive a pregnancy test. This is a standard test performed in the ED and considered part of routine practice. A pregnancy test in females is one test that is required by all patients undergoing this clearance among other labs not applicable to this study.

Baseline pain score will be determined using a 100 mm visual analogue scale, described to the patient as "no pain" being 0 and "the worst pain imaginable" being 100. A patient will be determined as eligible for enrollment if a baseline VAS score of 50 or greater is reported. A study investigator will then record the patient's body weight and baseline vital signs. Additional demographics recorded will include age, gender, comorbid medical conditions and headache classification.

Once the subject is determined to meet the inclusion/exclusive criteria and has agreed to participate in the study and has a signed consent form, the patient will be randomized via permutated-block randomization into the ketamine or standard care treatment group. An intravenous catheter will be initiated in each subject and 1000 mL normal saline IV bag will started on each patient per provider discretion.62 Once the medication of either treatment arm has been obtained and is ready to administer the PI or AI will document time zero.

The standard care arm will be administered 10mg of MET, 25 mg of DIP and +/- 15-30 mg of KET and +/- 10mg of dexamethasone IV push. 10 mg of MET will be added to the 1000 mL normal saline bag and infused as a bolus until the 1000 mL normal saline bag is empty. In addition, the standard care arm will be administered same volume of atomized intranasal normal saline as calculated dose of 0.75mg/kg ketamine.

The Ketamine arm will be administered intranasal SDDK via atomizer based on previous studies regarding intranasal ketamine administration in the ED at an initial dose of 0.75 mg/kg.2 The treating nurse will prepare the SDDK using the weight based dosing table found in each study packet. The treating nurse will give the syringe with the SDDK to the AI/PI for verification and administration. Each patient will also be administered 0.5ml, 0.5-1ml and 2.5ml normal saline boluses in place of the DIP, +/- KET and +/- DEX for a maximum of three boluses. An additional 2ml normal saline bolus will be added to the 1000 mL normal saline bag in place of the MET and the 1000 mL normal saline bag will be infused as a bolus until the bag is empty. Approximately 30 minutes after initial ketamine administration, study subjects will be asked if they would like an additional dose of medication for their headache. If the study subject request additional medication, the patient can receive a single repeat dose of 0.25mg/kg intranasal ketamine . This time was chosen empirically as reasonable time frame for clinic reassessment of analgesic affect.

60 minutes after all medications are given, subject participation in the study will be concluded and routine ED care will be resumed. At this time each subject will be asked if they would like additional medication for the treatment of their headache. If they would like additional medication, rescue analgesia may be given at the discretion of the ED provider managing the patient. Also, at any point the treating provider feels analgesia is inadequate either by patient verbalization or provider assessment, rescue medications may be provided at the treating provider's discretion.

Study investigators will record treatment arm pain scores, vital signs, and adverse effects at 10, 30, 60 and 90 minutes. Total hospital course time will also be documented. Adverse effects recorded will be based on the Side Effects Rating Scale for Dissociative Anesthetics (SERDA) and will include fatigue, dizziness, nausea, headache, feelings of unreality, changes in hearing, mood change, general discomfort and hallucinations. Although SERDA is frequently reported on a five point scale, patients will be graded on the adverse effects by answering "yes" or "no". An adverse effect will be considered serious if they resulted in clinical symptoms that were unable to be abated with clinical intervention or the tincture of time.

At the time of discharge, a final pain score will be recorded using the 10 point numerical rating score (NRS) with 0 meaning 'no pain' and 10 meaning "the worse pain possible." Patients will also be asked if they believed they got the study drug or standard care. A final ED encounter satisfaction score will be recorded using a the 10 point numerical rating score (NRS) with 0 meaning ' Very dissatisfied' and 1-0 meaning "Very satisfied." Follow-up will occur via telephone using the scripted phone conversation (included in this package) at 48-72 hours post-discharge. All subjects will be queried via a scripted interview for any adverse effects using the SERDA elements and whether the patient continues to perceive headache pain and duration of previous headache relief. Again, pain will be assessed using the 10 point NRS. Additional information will be collected via follow up communication including, but not limited to changes in medications, new diagnoses, unplanned visits or admissions.

Subject will be asked for contact information including phone numbers and email addresses for follow-up. Phone contact will be the primary method of contact. If, after two phone call attempts, the PI is unsuccessful at establishing patient contact, a scripted email be sent requesting the subject contact the protocol staff to complete the survey. If patients are unable to be contacted or lost to follow-up medical records will be queried for additional contact phone numbers if available. Veteran's Affairs system will be searched if all other methods are exhausted without result. The protocol team will attempt to contact the patient for 5 days after their hospital discharge date. If the patient has not been contacted by this time frame subjects will assumed to be lost to follow-up.

The primary outcome will be the change in pain level as documented by the VAS from study initiation to discharge. Secondary outcomes will include treatment efficiency (time to pain relief), change of pain score from discharge to follow up and side effects profile using the SERDSA questionnaire. All research will be completed when either the PI or AI are available in the ED to enroll and consent patients.

ELIGIBILITY:
Inclusion Criteria:

1. Chief compliant of a benign, non-life threatening headache that the PI/AI believe will require parental analgesia for management.
2. Ability to comprehend, speak, read, and write in the English language

Exclusion Criteria:

1. Age less than 18 and greater than 65
2. History of hypersensitivity to Ketamine, diphenhydramine, metoclopramide, ketorolac or dexamethasone
3. Weight less than 45 kg or more than 115 kg
4. Pregnancy or lactating female.
5. Patient is female of child-bearing age and unwilling to provide urine or blood for HCG analysis
6. Altered mental, diminished decision making capacity
7. Poor vital sign stability Hypoxia: O2 < 92%, Hypotension: SBP< 80 Hypertension: SBP>220 Heart rate: < 50 or >150 Respiratory Rate: <8 or >30
8. Presence of chronic oxygen-dependent pulmonary disease, liver cirrhosis, or renal disease requiring dialysis
9. Presence of ischemic heart disease, heart failure, or a history of unstable dysrhythmias
10. History of schizophrenia, psychosis or hallucinations (as assessed by electronic chart review)
11. History of alcohol or drug abuse
12. History of intracranial hypertension
13. History of glaucoma
14. History of HIV or immunosuppression
15. Presence of intracranial mass or vascular lesion (defined as inclusion criteria 1. As benign headaches)
16. Poorly controlled thyroid disease
17. Concomitant infections
18. History of pheochromocytoma
19. History of epilepsy
20. History of active bleeding or those receiving anticoagulants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
VAS 30 min | 30 min
  Change in Visual Analogue Score at 30 minutes

SECONDARY OUTCOMES:
VAS 60 min | 60 min
  Change in Visual Analogue Score at 60 minutes
NRS at discharge | Discharge
  Numerical Rating Scale at discharge
NRS 24 hours | 24 hours
  Pain NRS score at 24 hours post discharge
NRS 72 Hours | 72 Hours
  Pain NRS score at 72 hours post discharge
Side effects | At 15 min then at 30 min intervals while in the ED
  Side effects reported by patients in both treatments arms
Repeat ED/primary care encounters | 24 and 72 hours
  Need for repeat patient evaluation at 24-72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No